CLINICAL TRIAL: NCT01995019
Title: PhaseIV Study of Intra-articular Methylprednisolone in TMJ Arthralgia
Brief Title: Arthralgia of the Temporomandibular Joint. Pain Relief Following One Intra-articular Injection of Methylprednisolone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Artralgia1; 2013-003365-34 (EudraCT Number)
Record Dates: First submitted 2013-11-20; First posted 2013-11-26 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Arthralgia; TMJ
Keywords: Arthralgia; Temporomandibular joint; corticosteroids; injection; intra-articular
MeSH Terms: conditions — Arthralgia | interventions — Methylprednisolone; Methylprednisolone Acetate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physiologic saline (Placebo Comparator): Sodium chloride 9 mg/ml liquid for parental use
  Interventions: Drug: Methylprednisolone
- Methylprednisolone (Experimental): Depo-Medrol 40 mg/ml, single dose, injection, intra-articular
  Interventions: Drug: Physiologic saline

INTERVENTIONS:
Drug: Methylprednisolone — 1 ml single dose Intra-articular Depo-Medrol 40 mg/ml
  Other Names: Depo-Medrol 40 mg/ml
  Arms: Physiologic saline
Drug: Physiologic saline — 1 ml intra-articular placebo
  Other Names: Sham substance
  Arms: Methylprednisolone

SUMMARY:
The hypothesis is that a single dose intra-articular injection of corticosteroids are effective in relieving temporomandibular arthralgia pain.

The purpose of the study is therefore to evaluate the effect of a single dose intra-articular methylprednisolone vs. placebo in a month perspective on subjects with unilateral arthralgia of the TMJ.

DETAILED DESCRIPTION:
This is a randomized blinded multicenter controlled study on 64 subjects (18 years or older) with the diagnosis of unilateral arthralgia of the TMJ.

The subject visit the clinic at three occasions; one enrollment visit, one baseline treatment visit and one evaluation visit one month after baseline.

One week after baseline a follow-up telephone call is made with the purpose to track adverse events.

Pain questionaries are completed morning, lunch and dinnertime during three days before treatment, five days after treatment and three days proceeding the evaluation visit.

The study ís planned to commence 10th December 2013 and last patient out 15th January 2015.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or above
* the diagnosis arthralgia in one TMJ
* understands Swedish both verbally and in written
* signed informed concent

Exclusion Criteria:

* TMJ sounds in terms of clicking (crepitation allowed))
* polyarthritis/connective tissue disease
* bilateral TMJ arthralgia
* fibromyalgia or other generalized pain
* ongoing infection
* ongoing dental treatment
* intra-articular corticosteroid injection of a TMJ the past 6 months
* previous surgery of the affected TMJ
* complex psychiatric/psychologic status
* institutionalized living including prisoners
* staff at the investigational clinic
* hypersensitive to local anesthetics
* hypersensitive to methylprednisolone
* hemophilia
* methemoglobinemia
* nursing
* compromized health status according to the judgment of the investigator
* concommitant use of the drugs cyclosporine, erythromycin, pentobarbital, itraconazole, ketoconazole, Rifampicin, Acetylsalicylic acid, Oral anticoagulant
* mentally retarded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2013-12-10 (Actual); Primary Completion 2017-03-15 (Actual); Study Completion 2017-03-15 (Actual)

PRIMARY OUTCOMES:
VAS pain score change at maximal mouth opening | 4 weeks
  100 mm analog Visual Analog Scale with endpoints "No pain" and "Worst pain imaginable" The intra-individual change of the VAS pain score between baseline and end of study

SECONDARY OUTCOMES:
VAS pain score change at jaw rest | 4 weeks
  100 mm analog Visual Analog Scale with endpoints "No pain" and "Worst pain imaginable" The intra-individual change of the VAS pain score between baseline and end of study
Instrument measures | 4 weeks
  JFLS GCPS PHQ-9 PGIC
Adverse events | 4 weeks
  Spontaneously reported by the subject or observed by the study staff from the baseline visit until the evaluation visit.
  Reported by the subject in response to open questioning at visits/phone calls from the baseline visit until the evaluation visit "Have you had any health problems since your last visit/contact?"

CONTACTS AND LOCATIONS:
Overall Officials: Göran Isacsson, DDS, Principal Investigator — Orofacial pain unit, Västmanland Hospital Västerås
Locations (7):
- Sweden (7):
  - Orofacial pain unit, Malar Hospital Eskilstuna, Eskilstuna, Södermanland County
  - Dental specialist clinic Kaniken, Uppsala, Uppland
  - Specialist clinic Stomatognathic physiology, Gothenburg, VastraGotaland
  - Specialist center, Uddevalla, VastraGotaland
  - Orofacial pain unit, Västmanland Hospital Västerås, Västerås, Västmanland County
  - Orofacial pain unit, Dental Specialist Education Center, Örebro
  - Orofacial pain unit Eastman Institute, Stockholm